CLINICAL TRIAL: NCT02683512
Title: GBE Deficiency (GSD IV and APBD) Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00060753
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Glycogen Storage Disease Type IV; Adult Polyglucosan Body Disease; GSD4; GSD IV; APBD
MeSH Terms: conditions — Glycogen Storage Disease Type IV; Polyglucosan Body Disease, Adult Form

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This is an observational study that consists of data abstraction from patient medical records.

SUMMARY:
Collection and review of clinical information related to glycogen branching enzyme (GBE) deficiency, diagnosed as Glycogen Storage Disease Type IV (GSD IV) or Adult Polyglucosan Body Disease (APBD generated during clinic visits.

DETAILED DESCRIPTION:
This natural history study will serve as a repository of clinical, laboratory, and biochemical information on individuals with GBE deficiency, diagnosed as either GSD IV or APBD. This information will allow a more definitive description of GBE deficiency to be developed, which will permit development of treatment strategies for this disease.

Duke will be the only site where this study takes place. However, since this is a rare disorder, participants who receive care for GBE deficiency at other institutions will be included. We will collect retrospective data from patient charts on diagnosed individuals, as far back as necessary to capture the clinical course of the disorder. Prospective data collected from patient charts after enrollment will be captured as well. Participant's medical records will be continually reviewed for the duration of the study.

Data will be collected from medical records and will only pertain to clinically relevant information, including, but not limited to: demographic and diagnostic information, tissue biopsy results, medical and family history, review of systems, imaging studies, results of liver, muscle, and nerve function testing, and urine and blood laboratory results.

ELIGIBILITY:
* Diagnosis of GSD IV or APBD via:

  * Two variants in the GBE1 gene
  * Deficient GBE activity in liver, muscle, skin fibroblast or other tissue
  * One variant in GBE1 gene with evidence of disease that is pathogenic, per the clinician
* Able to provide informed consent for self (adults) or affected individual (minor or adults with a legally authorized representative)
* Able to provide consent for release of medical records
* Pregnant women with a diagnosis of GSD IV or APBD will be included
* Histology as confirmed by clinician

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with GBE deficiency, diagnosed as GSD IV or APBD, regardless of gender or ethnicity, are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Progression of disease | Duration of study, approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koch RL, Kiely BT, Choi SJ, Jeck WR, Flores LS, Sood V, Alam S, Porta G, LaVecchio K, Soler-Alfonso C, Kishnani PS. Natural history study of hepatic glycogen storage disease type IV and comparison to Gbe1ys/ys model. JCI Insight. 2024 May 14;9(12):e177722. doi: 10.1172/jci.insight.177722. PMID 38912588